CLINICAL TRIAL: NCT03658889
Title: Cross-sectional, Multicentre, Non-interventional Study to Assess Giant Cell Arteritis Medical Practices in France
Brief Title: Assessment of Giant Cell Arteritis Medical Practices in France
Acronym: ARTEMIS
Status: Completed | Type: Observational
Sponsor: Chugai Pharma France (Industry)
Collaborators: ITEC Services (Other)
Responsible Party: Sponsor
Other Study IDs: CPF_ARTEMIS2018
Record Dates: First submitted 2018-07-11; First posted 2018-09-06 (Actual); Results first posted 2020-05-28 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients under treatment(s) for GCA: Patients at least 50 years old with Giant Cell Arteritis (GCA) and under treatment(s) for GCA

SUMMARY:
The purpose of this study is to describe medical practices in patients with GCA in terms of patient journey, diagnostic methods and specific GCA treatments since diagnosis.

DETAILED DESCRIPTION:
This is a cross-sectional, non-interventional, national (France), multicentre study, conducted on a population of 300 patients with GCA, to describe GCA management and patient characteristics.

The study will be conducted in accordance with the professional code of ethics and the good epidemiological practice guidelines developed by the Association of French-Speaking Epidemiologists.

The information will be collected during a single visit to the internist or rheumatologist as part of the usual management of the patient with GCA. The physician will not perform any additional examinations specific to the study. The physician will inform the patient about the study before inclusion and seek her/his non-opposition. A patient information form will be given to each patient by the physician. Patients who are eligible to participate in the study and who verbally accept automatic processing of their personal data, will be included in the study.

Data will be collected from the medical file and from patient questionnaires on health status (SF-36 [36-Item Short Form Survey Instrument], EQ5D [EuroQol-5 Dimensions]) and fatigue (FACIT-fatigue). In addition, GCA activity will be evaluated using a global arteritis activity Visual Analog Scale (VAS) to be completed by the patient and the physician.

ELIGIBILITY:
Inclusion Criteria:

* At least 50 years old.
* Suffering from GCA as per investigator judgement, newly diagnosed or not.
* Starting or under treatment for GCA.
* Informed verbally and in writing about this study and not objecting to their data being electronically processed or subjected to data quality control.

Non-inclusion Criteria:

* Unable to consent
* Participation to a randomised controlled clinical trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 patients aged at least 50 years old, suffering from GCA, starting or under treatment for GCA recruited by 150 internists and rheumatologists practicing in hospitals or private clinics in Metropolitan France will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred MAHR, Professor, Principal Investigator — alfred.mahr@aphp.fr
Locations (1):
- Hospital of the Archet, Nice, Alpes-Maritimes, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Physicians: Physicians who recruited the patients with Giant Cell Arteritis (GCA)
Period: Overall Study
Arm/Group | Patients Under Treatment(s) for GCA | Physicians
Started | 308 (Enrolled population) | 69
Completed | 306 (Analysis population) | 69
Not Completed | 2 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Under Treatment(s) for GCA | Physicians | Total
Number analyzed (Participants) | 306 | 69 | 375
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Physician age was not collected
  years
    number analyzed (Participants) | 306 | 0 | 306
    (all) | 73.98 (7.88) |  | 73.98 (7.88)
Age, Customized [Count of Participants; unit: Participants] — Population: Physician age was not collected
  Participants
    [50-70[ years: number analyzed (Participants) | 306 | 0 | 306
    [50-70[ years | 84 |  | 84
    ≥ 70 years: number analyzed (Participants) | 306 | 0 | 306
    ≥ 70 years | 222 |  | 222
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206 | 21 | 227
  Male | 100 | 48 | 148
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Physician who follows the patient [Count of Participants; unit: Participants] — Population: This measure is not relevant for the physician population
  Participants
    number analyzed (Participants) | 306 | 0 | 306
    Internal Medicine | 258 |  | 258
    Rheumatologist | 46 |  | 46
    Geriatry | 2 |  | 2
Patients' medical history [Count of Participants; unit: Participants] — The most frequent SOCs (>10% of patients) of events occurring before GCA diagnosis Population: this measure is not relevant for the physician population
  Participants
    Vascular disorders: number analyzed (Participants) | 306 | 0 | 306
    Vascular disorders | 148 |  | 148
    Metabolism and nutrition disorders: number analyzed (Participants) | 306 | 0 | 306
    Metabolism and nutrition disorders | 73 |  | 73
    Musculoskeletal and connective tissue disorders: number analyzed (Participants) | 306 | 0 | 306
    Musculoskeletal and connective tissue disorders | 52 |  | 52
    Cardiac disorders: number analyzed (Participants) | 306 | 0 | 306
    Cardiac disorders | 41 |  | 41
    Eye disorders: number analyzed (Participants) | 306 | 0 | 306
    Eye disorders | 40 |  | 40
    Psychiatric disorders: number analyzed (Participants) | 306 | 0 | 306
    Psychiatric disorders | 31 |  | 31
Patients' comorbidities [Count of Participants; unit: Participants] — The most frequent SOCs (>10% of patients) of events with ongoing specific treatments Population: This measure is not relevant for the physician population
  Participants
    Vascular disorders: number analyzed (Participants) | 306 | 0 | 306
    Vascular disorders | 140 |  | 140
    Metabolism and nutrition disorders: number analyzed (Participants) | 306 | 0 | 306
    Metabolism and nutrition disorders | 79 |  | 79
    Musculoskeletal and connective tissue disorders: number analyzed (Participants) | 306 | 0 | 306
    Musculoskeletal and connective tissue disorders | 43 |  | 43
    Cardiac disorders: number analyzed (Participants) | 306 | 0 | 306
    Cardiac disorders | 41 |  | 41
    Psychiatric disorders: number analyzed (Participants) | 306 | 0 | 306
    Psychiatric disorders | 37 |  | 37
Treatments concomitant to diagnosis [Count of Participants; unit: Participants] — Number of patients taking at least one of the following treatments at diagnosis Population: Analysis population for whom the data is not missing
  Participants
    Antiplatelets: number analyzed (Participants) | 304 | 0 | 304
    Antiplatelets | 68 |  | 68
    Statins: number analyzed (Participants) | 305 | 0 | 305
    Statins | 40 |  | 40
    Antiosteoporotics: number analyzed (Participants) | 304 | 0 | 304
    Antiosteoporotics | 26 |  | 26
    Antihypertensives: number analyzed (Participants) | 305 | 0 | 305
    Antihypertensives | 141 |  | 141
    Antidiabetics: number analyzed (Participants) | 304 | 0 | 304
    Antidiabetics | 25 |  | 25
    Inhibitors of the proton pump: number analyzed (Participants) | 305 | 0 | 305
    Inhibitors of the proton pump | 67 |  | 67
    Hypnotics: number analyzed (Participants) | 305 | 0 | 305
    Hypnotics | 29 |  | 29
    Antidepressants: number analyzed (Participants) | 306 | 0 | 306
    Antidepressants | 22 |  | 22
    CA Vit D: number analyzed (Participants) | 306 | 0 | 306
    CA Vit D | 22 |  | 22
    Other: number analyzed (Participants) | 305 | 0 | 305
    Other | 53 |  | 53
Treatments concomitant to inclusion [Count of Participants; unit: Participants] — Number of patients taking at least one of the following treatments at inclusion Population: Analysis population for whom the data is not missing
  Participants
    Antiplatelets: number analyzed (Participants) | 305 | 0 | 305
    Antiplatelets | 158 |  | 158
    Statins: number analyzed (Participants) | 304 | 0 | 304
    Statins | 64 |  | 64
    Antiosteoporotics: number analyzed (Participants) | 304 | 0 | 304
    Antiosteoporotics | 112 |  | 112
    Antihypertensives: number analyzed (Participants) | 304 | 0 | 304
    Antihypertensives | 152 |  | 152
    Antidiabetics: number analyzed (Participants) | 304 | 0 | 304
    Antidiabetics | 48 |  | 48
    Inhibitors of the proton pump: number analyzed (Participants) | 305 | 0 | 305
    Inhibitors of the proton pump | 130 |  | 130
    Hypnotics: number analyzed (Participants) | 305 | 0 | 305
    Hypnotics | 35 |  | 35
    Antidepressants: number analyzed (Participants) | 305 | 0 | 305
    Antidepressants | 31 |  | 31
    CA Vit D: number analyzed (Participants) | 306 | 0 | 306
    CA Vit D | 70 |  | 70
    Other: number analyzed (Participants) | 305 | 0 | 305
    Other | 79 |  | 79

OUTCOME MEASURES:

1. Primary Outcome: Patient Journey : Physicians Who Referred the Patient
Description: Proportion of patients for each physician specialty that referred the patient
Time Frame: Baseline only
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 306
Participants
  General Practitioner | 171
  Ophthalmologist | 31
  Neurologist | 21
  Emergency | 17
  Internist | 13
  Rheumatologist | 15
  Other | 12
  Anatomical Pathologist | 0
  Angiologist/Vascular doctor | 7
  Cardiologist | 10
  Surgeon/Vascular surgeon | 3
  Endocrinologist/Diabetologist | 1
  Gastro-enterologist | 0
  Geriatrician | 3
  Ear, Nose and Throat specialist (ENT) | 0
  Pulmonologist | 1
  Radiologist | 1

2. Primary Outcome: Patient Journey : Physician Encountered by the Patient at Least One Time Since the First Events Related to GCA
Description: Physician encountered by the patient at least one time since the first events related to GCA (Multiple answers possible, If a patient encountered a medical speciality more than one time, this speciality will be counted only once)
Time Frame: Baseline only
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 306
Participants
  General Practitioner | 260
  Ophthalmologist | 88
  Neurologist | 38
  Emergency | 54
  Internist | 59
  Rheumatologist | 42
  Anatomical pathologist | 3
  Angiologist/Vascular surgeon | 17
  Cardiologist | 20
  Surgeon/Vascular surgeon | 9
  Endocrinologist/Diabetologist | 3
  Gastro-enterologist | 6
  Geriatrician | 3
  Ear, Nose, Throat specialist (ENT) | 9
  Pulmonologist | 5
  Radiologist | 7
  Other | 30

3. Primary Outcome: Patient Journey : Time to GCA Diagnosis
Description: Time between GCA signs/symptoms and diagnosis
Time Frame: Baseline only
Population: Analysis population (missing data for 2 patients)
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 304
months | 1.00 [1.00 to 3.00]

4. Primary Outcome: GCA Diagnostic Method
Description: Proportions of each diagnostic method used
Time Frame: Baseline only
Population: Patients for whom the data is filled (ESR, n=285; C-Reactive Protein [CRP], n=275; Temporal Artery Biopsy [TAB], n=294; High resolution echo Doppler, n=292; MRI of the temporal arteries, n=304; 18 Fluorodeoxyglucose-positron emission tomography [18FDG-PET], n=280; Aortic angio-CT, n=293)
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 306
Participants
  Erythrocyte Sedimentation Rate (ESR: number analyzed (Participants) | 285
  Erythrocyte Sedimentation Rate (ESR | 154
  C-Reactive Protein (CRP): number analyzed (Participants) | 275
  C-Reactive Protein (CRP) | 266
  Biopsy of the Temporal Artery (TAB): number analyzed (Participants) | 294
  Biopsy of the Temporal Artery (TAB) | 249
  High resolution color Doppler ultrasound: number analyzed (Participants) | 292
  High resolution color Doppler ultrasound | 91
  MRI of the temporal arteries: number analyzed (Participants) | 304
  MRI of the temporal arteries | 20
  18FDG PET: number analyzed (Participants) | 280
  18FDG PET | 74
  Aortic angio-CT: number analyzed (Participants) | 293
  Aortic angio-CT | 87

5. Primary Outcome: GCA Treatments Since Diagnosis : Glucocorticoids Since Diagnosis
Description: GCs treatment since diagnosis : Current GC dose at inclusion and total cumulative GC dose according to investigator (excl. IV bolus) since diagnosis.
Time Frame: Baseline only
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 306
mg
  Current dose at inclusion | 9.00 [5.00 to 20.00]
  Total cumulative dose | 4305.00 [1920.00 to 7000.00]

6. Primary Outcome: GCA Treatments Since Diagnosis: Glucocorticoids at Inclusion
Description: Number of patients with at least one GC kinetic ongoing at inclusion
Time Frame: baseline only
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 306
Participants | 273

7. Primary Outcome: GCA Treatments Since Diagnosis: Immunosuppressants Stopped Before Inclusion
Description: Immunosuppressants for GCA taken since diagnosis and stopped before inclusion
Time Frame: Baseline only
Population: among analysis population, 27 patients have taken at least one immunosuppressant since diagnosis and stopped before inclusion
Measure: Number; unit: number of treatments
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 27
number of treatments
  Azathioprine | 2
  Cyclophosphamide | 1
  Cyclosporine | 0
  Leflunomide | 1
  Methotrexate | 25
  Mycophenolate Mofetil | 0
  Other | 0

8. Primary Outcome: GCA Treatments Since Diagnosis: Immunosuppressants Ongoing at Inclusion
Description: Number of patients with at least one immunosuppressant ongoing at inclusion
Time Frame: Baseline only
Population: Among analysis population, 35 Patient had at least one immunosuppressant ongoing at inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 35
Participants
  Azathioprine | 0
  Cyclophosphamide | 0
  Cyclosporine | 0
  Leflunomide | 0
  Methotrexate | 35
  Mycophenolate Mofetil | 0
  Other | 0

9. Primary Outcome: GCA Treatments Since Diagnosis: Targeted Biologic Therapies Stopped Before Inclusion
Description: Number of patients who have taken at least one targeted biologic therapy since diagnosis and stopped before inclusion
Time Frame: Baseline only
Population: Among analysis population, 8 patients have taken at least one targeted biologic therapy since diagnosis and stopped before inclusion
Measure: Number; unit: treatments
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 8
treatments
  Adalimumab | 1
  Abatacept | 0
  Etanercept | 0
  Infliximab | 0
  Tocilizumab | 9
  Other | 0

10. Primary Outcome: GCA Treatments Since Diagnosis: Targeted Biologic Therapies Ongoing at Inclusion
Description: Number of patients with at least one targeted biologic therapy ongoing at inclusion
Time Frame: Baseline only
Population: Among analysis population, 45 patients had at least one targeted biologic therapy ongoing at inclusion
Measure: Number; unit: treatments
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 45
treatments
  Adalimumab | 0
  Abatacept | 0
  Etanercept | 0
  Infliximab | 1
  Tocilizumab | 44
  Other | 0

11. Secondary Outcome: Comorbidities Related to GCs
Description: Comorbidities related/ aggravated by the use of GCs according to the investigator's judgment in at least 2 patients (by SOC)
Time Frame: Baseline only
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 306
Participants
  Cardiac disorders | 5
  Endocrine disorders | 2
  Eye disorders | 9
  Gastrointestinal disorders | 4
  Hepatobiliary disorders | 2
  Infections and infestations | 10
  Injury, poisoning and procedural complications | 7
  Investigations | 4
  Metabolism and nutrition disorders | 44
  Musculoskeletal and connective tissue disorders | 25
  Nervous system disorders | 7
  Psychiatric disorders | 18
  Renal and urinary disorders | 2
  Respiratory, thoracic and mediastinal disorders | 3
  Surgical and medical procedures | 4
  Vascular disorders | 33

12. Secondary Outcome: Treatments in Patients With Comorbidities Related to GCs
Description: Number of patients with at least one ongoing treatment for comorbidities related to the use of GCs
Time Frame: Baseline only
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 306
Participants | 98

13. Secondary Outcome: Proportion of Incident Patients
Description: Proportion of incident patients: patients with a diagnosis of GCA ≤ 6 weeks from inclusion
Time Frame: Baseline only
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 306
Participants | 39

14. Secondary Outcome: Proportion of Prevalent Patients
Description: Proportion of prevalent patients: patients with a diagnosis of GCA > 6 weeks from inclusion
Time Frame: Baseline only
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 306
Participants | 267

15. Secondary Outcome: GCA Duration
Description: Time since GCA diagnosis for overall population, prevalent and incident patients
Time Frame: Baseline only
Population: Overall analysis population: N=306 / Prevalent patients (GCA diagnosis>6weeks), N=267 / Incident patients (GCA diagnosis ≤ 6weeks), N=39
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 306
months
  Overall population | 13.00 [5.00 to 26.00]
  Prevalent patients: number analyzed (Participants) | 267
  Prevalent patients | 15.00 [7.00 to 30.00]
  Incident patients: number analyzed (Participants) | 39
  Incident patients | 0.60 [0.20 to 1.00]

16. Secondary Outcome: GCA Initial Presentation
Description: Proportions of patients with cranial GCA, Polymyalgia Rheumatica (PMR), extracranial GCA, elevated ESR/CRP and general signs at diagnosis
Time Frame: Baseline only
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 306
Participants
  at least one cranial manifestation | 271
  at least one PMR symptom | 148
  at least one extracranial event (excl. PMR) | 108
  Value of ESR (mm/1st h) > 50 mm/h | 129
  at least one general sign | 227

17. Secondary Outcome: GCA Clinical Form
Description: Proportion of patients with at least one relapse and number of relapses
Time Frame: Baseline only
Population: Prevalent patients
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 267
Participants
  Patients with 1 relapse | 69
  Patients with 2 relapses | 32
  Patients with 3 relapses | 11
  Patients with 4 relapses | 6
  Patients with 5 relapses | 4

18. Secondary Outcome: Patients With GCA Complications
Description: Proportions of patients with GCA complications
Time Frame: Baseline only
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 306
Participants | 48

19. Secondary Outcome: Global Arteritis Activity
Description: Score of the physician and patient global arteritis activity on a 100 mm-visual analog scale (100mm-VAS) (Patients with physician's VAS score less than or equal to 10mm will be considered with "non-active GCA", while patients with physician's VAS score greater than 10 mm will be considered with "active GCA")
Time Frame: Baseline only
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 306
mm
  Patient VAS score | 18.00 [5.00 to 47.00]
  Physician VAS score | 4.00 [1.00 to 14.00]

20. Secondary Outcome: Patient Reported Outcome (PRO) Scores: Short Form-36 (SF-36) Questionnaire
Description: Total and detailed scores of the self reported SF-36 questionnaire (36-Item Short Form Survey Instrument): 36 item survey measuring health-related quality-of-life.
  For each domains: score ranging from 0 (worst health status) to 100 (best health status)
Time Frame: Baseline only
Population: Analysis population, SF-36 scores were missing for 11 patients
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 295
mm
  Physical functioning: number analyzed (Participants) | 283
  Physical functioning | 70.00 [45.00 to 90.00]
  Physical role functioning: number analyzed (Participants) | 286
  Physical role functioning | 56.25 [31.25 to 87.50]
  Bodily pain: number analyzed (Participants) | 287
  Bodily pain | 62.00 [31.25 to 87.50]
  General health: number analyzed (Participants) | 288
  General health | 57.00 [42.00 to 72.00]
  Emotional role functioning: number analyzed (Participants) | 288
  Emotional role functioning | 66.67 [41.67 to 91.67]
  Vitality: number analyzed (Participants) | 285
  Vitality | 50.00 [31.25 to 68.75]
  Emotional well-being: number analyzed (Participants) | 287
  Emotional well-being | 60.00 [45.00 to 80.00]
  Social functioning: number analyzed (Participants) | 278
  Social functioning | 60.00 [45.00 to 80.00]
  Physical component summary (PCS): number analyzed (Participants) | 261
  Physical component summary (PCS) | 46.25 [38.35 to 52.81]
  Mental component summary (MCS): number analyzed (Participants) | 261
  Mental component summary (MCS) | 44.52 [34.43 to 53.06]

21. Secondary Outcome: PRO Scores: EQ5D-3L Questionnaire
Description: Total score of the EuroQol-5 Dimensions 3 Levels (EQ5D-3L) questionnaire and perceived current health state (100mm-EQ_VAS score, 0 = 'Worst imaginable health state' and 100 = 'Best imaginable health state)
Time Frame: Baseline only
Population: Analysis population: 303 EQ-5D-3L questionnaires were completed
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 303
score on a scale
  EQ-5D-3L score: number analyzed (Participants) | 289
  EQ-5D-3L score | 0.79 [0.56 to 0.87]
  EQ_VAS score: number analyzed (Participants) | 301
  EQ_VAS score | 69.00 [50.00 to 80.00]

22. Secondary Outcome: PRO Scores: FACIT-Fatigue Questionnaire
Description: Total score of the 13-items Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) questionnaire.
  FACIT-Fatigue is an instrument that measures overall fatigue and its effects on the general functioning and daily activities through 13 questions. Each question has 5 levels: not at all, a little bit, somewhat, quite a bit, very much. Lower scores indicate greater fatigue. The total score of FACIT-Fatigue varies from 0 to 52 (score <30 = severe fatigue).
Time Frame: Baseline only
Population: Analysis population: 300 patients completed the FACIT-fatigue questionnaire
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Patients Under Treatment(s) for GCA
Number analyzed (Participants) | 300
score on a scale | 39.00 [28.00 to 46.00]

23. Secondary Outcome: Physician Medical Specialty
Description: Physician characteristics: medical specialty
Time Frame: Baseline only
Measure: Count of Participants; unit: Participants
Groups:
- Physician Population: Physicians who recruited the patients with Giant Cell Arteritis (GCA)
Arm/Group | Physician Population
Number analyzed (Participants) | 69
Participants
  Internal Medicine | 56
  Rheumatology | 12
  Geriatry | 1

24. Secondary Outcome: Physician Number of Years of Practice
Description: Number of years since medical school graduation
Time Frame: Baseline only
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | Physician Population
Number analyzed (Participants) | 69
years | 13.00 [6.00 to 20.00]

25. Secondary Outcome: Physician Type of Practice
Description: Physician main activity (University Hospital or General Services Hospital)
Time Frame: Baseline only
Measure: Count of Participants; unit: Participants
Arm/Group | Physician Population
Number analyzed (Participants) | 69
Participants
  University Hospital | 39
  General Services Hospital | 30

26. Secondary Outcome: Physician Characteristics: Number of GCA Diagnosis
Description: Number of GCA cases (Horton) personally treated within the last year prior to the date of inclusion of first patient
Time Frame: Baseline only
Population: 1 physician for whom the data is missing
Measure: Count of Participants; unit: Participants
Arm/Group | Physician Population
Number analyzed (Participants) | 68
Participants
  1 to 2 cases | 2
  3 to 5 cases | 17
  6 to 10 cases | 12
  11 to 20 cases | 16
  more than 20 cases | 21

ADVERSE EVENTS:
Description: This was a descriptive observational study on GCA characteristics and management in a real-life setting with no specific medicinal product to be investigated. No adverse events and reactions were collected.
Arm/Group | Patients Under Treatment(s) for GCA
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT03658889/Prot_002.pdf
  • Statistical Analysis Plan (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT03658889/SAP_003.pdf